CLINICAL TRIAL: NCT07129889
Title: The Efficacy and Safety of Auricular Acupressure for Reducing the Rebound Phenomenon in Myopic Children After Discontinuing 0.01% Atropine Eye Drops: A Three-Arm, Blinded Randomized Controlled Trial Study Protocol
Brief Title: Auricular Acupressure Reduces Rebound Effects After Discontinuation of Atropine
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ningbo Eye Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ningbo Eye Hospital
Record Dates: First submitted 2025-08-07; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Myopia
Keywords: Auricular acupressure; myopia; atropine; rebound effect; randomized controlled trial
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- the atropine tapering group (Active Comparator): Patients were administered 0.01% atropine eye drops using a gradual reduction method (Shenyang Xingqi Eye Pharmaceutical Co., Ltd., Shenyang, China, National Medical Products Administration license number: H20243320, 0.04 mg) . The dose was reduced by one day each month, ultimately reducing atropine treatment from seven days per week to complete withdrawal within six months, with a six-month follow-up.
  Interventions: Drug: gradual withdrawal of medication
- Auricular acupressure (Experimental): AA therapy will be added to the gradual reduction method of 0.01% atropine eye drops. As shown in Figure 1. 2; Table 2, ear acupoints: Shenmen (TF4), Heart (CO15), Liver (CO12), Spleen (CO13), Kidney (CO10), and Eye (LO5). The acupuncturist first uses a metal probe to locate the ear acupoints and asks the patient if they feel "deqi," such as heat, numbness, swelling, or pain. After confirming the ear acupoints, the ears are cleaned with a 75% ethanol solution and dried with sterile, dry cotton balls. Subsequently, the acupuncturist uses the left hand to stabilize the ear while the right hand uses tweezers to apply adhesive tape (10 × 10 mm) containing Wangbuluxing seeds (Wujiang Jiacheng Acupuncture Instrument Co., Ltd., Suzhou, China) to the selected auricular regions.
  Interventions: Procedure: Auricular acupressure
- Sham Auricular acupressure (Sham Comparator): Acupuncturists will use a gradual reduction method with 0.01% atropine eye drops, as used in the control group, and apply skin-colored adhesive tape without Wang Bu Liu Xing seeds to the ear acupoints. During treatment, no massage or acupoint pressure will be applied. The SAA group will follow the same protocol as the AA group for compensatory AA treatment at the end of the study.
  Interventions: Procedure: Sham auricular acupressure

INTERVENTIONS:
Drug: gradual withdrawal of medication — The dose was reduced by one day each month, ultimately reducing atropine treatment from seven days per week to complete withdrawal within six months, with a six-month follow-up.
  Arms: the atropine tapering group
Procedure: Auricular acupressure — First, treat the ear acupoint on one side, then leave the tape in place for 5 days. On the 6th day, remove the tape, rest for 2 days, and on the 8th day, apply new tape to the other side of the ear. Changing the tape aims to minimize adverse event (AE) that may result from prolonged stimulation on one side. Additionally, participants will be instructed to self-administer vertical pressure on the Wangbuluxing seeds 15-20 times to achieve sensation, with a duration of 4-5 times daily. The treatment process will last for 18 months, with a follow-up at 6 months.
  Arms: Auricular acupressure
Procedure: Sham auricular acupressure — Acupuncturists will use a gradual reduction method with 0.01% atropine eye drops, as used in the control group, and apply skin-colored adhesive tape without Wang Bu Liu Xing seeds to the ear acupoints. During treatment, no massage or acupoint pressure will be applied. The SAA group will follow the same protocol as the AA group for compensatory AA treatment at the end of the study.
  Arms: Sham Auricular acupressure

SUMMARY:
0.01% atropine is an effective measure for controlling myopia in children and is widely used in Asia for this purpose. However, there is a phenomenon of rebound and worsening of myopia after discontinuation of the medication. Auricular acupressure (AA) is gaining attention as a complementary therapy for myopia control. However, there is a lack of rigorous studies evaluating the effectiveness of AA in reducing rebound after discontinuing atropine eye drops in myopic children. Our study aims to assess the efficacy and safety of AA in reducing rebound after discontinuing atropine in myopic children.

DETAILED DESCRIPTION:
This study is a randomized, single-blind, three-arm controlled trial. At least 180 participants will be randomly assigned to one of three groups: the atropine tapering group, the AA group, and the sham auricular acupressure (SAA) group. All treatments will be conducted over 1.5 years, with a 6-month follow-up. The primary outcome measure is the rate of myopia rebound. Secondary outcome measures include annual growth rate of spherical equivalent (SE), annual growth rate of axial length (AL), annual delay rate of SE, annual delay rate of AL, annual delay rate of SE, annual delay rate of AL, choroidal thickness (ChT), choroidal vascular index (CVI), and choroidal vascular volume (CVV). Intention-to-treat and per-protocol analyses will be conducted, with a significance level set at 5%.

ELIGIBILITY:
Inclusion Criteria:

1. Meets the diagnostic criteria for myopia;
2. Age 6-12 years, no gender restrictions;
3. Single or bilateral spherical refractive error between -1.00 and -4.00 D (astigmatism ≤ 1.50 D, anisometropia ≤ 1.50 D);
4. Best-corrected visual acuity in both eyes of 0.20 logMAR or higher;
5. Intraocular pressure (IOP) less than 21 mmHg;
6. Informed consent form signed by a guardian, voluntarily participating.

Exclusion Criteria:

Patients who meet any of the following criteria will not be eligible to participate in the study:

1. Eye conditions other than refractive errors (e.g., strabismus, amblyopia, keratitis, glaucoma, cataracts, retinal detachment, etc.);
2. Patients with systemic conditions that may affect refractive development (e.g., Down syndrome, Marfan syndrome);
3. Patients with uncontrolled systemic diseases or debilitating conditions, immune deficiencies, or severe primary diseases of the cardiovascular, hepatic, renal, or hematopoietic systems, immune system disorders, or psychiatric conditions;
4. Patients with a history of allergies or hypersensitivity to multiple medications;
5. Patients who have undergone ocular surgery within the past 4 weeks prior to screening;
6. Patients planning to undergo ocular surgery within one year of enrollment;
7. Patients who have participated in other drug clinical trials within the past 3 months prior to screening; Patients who are unable to cooperate with treatment, observation, and assessment.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2025-12-02 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Myopia Rebound Rate | Statistical analysis was performed at 3 months and 6 months after dose reduction, and at 1 month, 3 months, and 6 months after discontinuation of medication.
  The myopia rebound rate is defined as the ratio of the number of individuals experiencing myopia rebound to the total number of individuals in each group. The rebound effect is defined as the rate of myopia progression after discontinuation of treatment exceeding the rate observed during the treatment phase. The rebound effect is assessed based on changes in AL or SE. To enable direct comparison, all data were standardized to an annual rate (mm/y or D/y) by dividing the change in SE or AL by the duration of follow-up (y).
  Myopia relapse rate = number of relapses / total number of participants × 100%

SECONDARY OUTCOMES:
spherical equivalent annual growth(SEA) | The measurement method is the same as above, with three consecutive measurements taken and the average calculated. Measurements are taken at 3, 6, and 9 months after intervention, 3 and 6 months after dose reduction, and 1, 3, and 6 months after disconti
  SE annual growth is defined as the annualized amount of SE after ciliary muscle paralysis.
  SE annual growth = SE change value / follow-up duration (y)
Axial length annual growth(ALA) | Measurements are taken at 3 months, 6 months, 9 months, and 12 months after intervention, 3 months and 6 months after dose reduction, and 1 month, 3 m
  The annual growth rate of AL is the annualized value of AL.The measurement method involves taking five consecutive measurements and calculating the average value.
  Annual growth rate of AL = Change in AL value / Follow-up duration (y)
SE year delay amount | Measurements are taken at 3 months, 6 months, 9 months, and 12 months after intervention, 3 months and 6 months after dose reduction, and 1 month, 3 months, and 6 months after discontinuation of medication.
  The SE delay is defined as the difference between the annual change in SE in the AA group, SAA group, and atropine withdrawal group after ciliary muscle paralysis.
  SE delay = |control group SEA - experimental group SEA|
AL year delay amount | Measurements are taken at 3 months, 6 months, 9 months, and 12 months after intervention, 3 months and 6 months after dose reduction, and 1 month, 3 months, and 6 months after discontinuation of medication.
  The AL-year delay is defined as the difference between the AL-year change in the AA group, SAA group, and atropine gradual withdrawal group.
  AL-year delay = |control group ALA - experimental group ALA|
SE year delay rate | Measurements are taken at 6 months, and 12 months after intervention, 6 months after dose reduction, and 6 months after discontinuation of medication.
  The SE annual delay rate is defined as the ratio of the SE annual delay amount to the SE annual change amount in the control group multiplied by 100%.
  SE annual delay rate = SE annual delay amount / SE annual change amount in the control group * 100%
AL year delay rate | Measurements are taken at 6 months, and 12 months after intervention, 6 months after dose reduction, and 6 months after discontinuation of medication.
  The AL annual delay rate is defined as the ratio of the AL annual delay amount to the AL annual change amount in the control group multiplied by 100%.
  AL annual delay rate = AL annual delay amount / AL annual change amount in the control group * 100%
choroidal thickness (ChT) | Measurements were taken at the start of the trial, 3, 6, 9, and 12 months after the intervention, 3 and 6 months after dose reduction, and 1, 3, and 6 months after discontinuation of medication.
  The Sub-Surface Optical Coherence Tomography Angiography (SS-OCTA) system employs Deep Layer™ artificial intelligence for layered measurement of choroidal thickness. Choroidal thickness measurement in the macular region: The macular region of the examined eye is designated as the scanning area, with the fovea centralis as the center, and a radial scan is performed in an ETDRS concentric circle pattern. Choroidal thickness is automatically calculated by the system. In the magnified OCTA image, measurements are taken below the fovea centralis, with nine regions-temporal, nasal, superior, inferior, superior temporal, inferior nasal, inferior temporal, and superior nasal-within the 0-3mm, 0-6mm, and 0-9mm ranges of the macula. The system automatically calculates the average choroidal thickness across the three ranges.
choroidal vascular index (CVI) | Measurements were taken at the start of the trial, 3, 6, 9, and 12 months after the intervention, 3 and 6 months after dose reduction, and 1, 3, and 6 months after discontinuation of medication.
  The measurement method for choroidal thickness and choroidal vascular volume uses B-scan mode, with a 9.00 × 9.00 mm vascular OCT scan centered on the fovea of each eye. The system automatically identifies the choroidal vascular structure, reconstructs the choroidal vascular morphology, and quantifies the choroidal vascular volume and vascular index. The vascular index and vascular index within the ETDRS ring range of 0-3 mm, 0-6 mm, and 0-9 mm are measured.
choroidal vascular volume (CVV) | Measurements were taken at the start of the trial, 3, 6, 9, and 12 months after the intervention, 3 and 6 months after dose reduction, and 1, 3, and 6 months after discontinuation of medication.
  The measurement method for choroidal thickness and choroidal vascular volume uses B-scan mode, with a 9.00 × 9.00 mm vascular OCT scan centered on the fovea of each eye. The system automatically identifies the choroidal vascular structure, reconstructs the choroidal vascular morphology, and quantifies the choroidal vascular volume and vascular index. The vascular index and vascular index within the ETDRS ring range of 0-3 mm, 0-6 mm, and 0-9 mm are measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Ningbo Eye Hospital, Ningbo, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2024-11-06): https://cdn.clinicaltrials.gov/large-docs/89/NCT07129889/Prot_SAP_000.pdf
  • Informed Consent Form: Parental Consent Form (2024-07-04): https://cdn.clinicaltrials.gov/large-docs/89/NCT07129889/ICF_001.pdf
  • Informed Consent Form: Informed Consent Form for Children (2024-07-04): https://cdn.clinicaltrials.gov/large-docs/89/NCT07129889/ICF_002.pdf